CLINICAL TRIAL: NCT05815641
Title: Analysis of the Pre- and Post-prandial Levels of Appetite Regulatory Hormones in Adult Individuals
Brief Title: Pre- and Post-prandial Levels of Appetite Regulatory Hormones in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020/0044
Record Dates: First submitted 2023-02-16; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Appetitive Behavior
MeSH Terms: conditions — Obesity; Appetitive Behavior | interventions — Food; Breakfast

STUDY DESIGN:
Intervention Model Description: Participants will be given a test meal (breakfast) that provides 20% of the individual's daily energy requirement. The breakfast composition is 56 kcal% carbohydrates, 12 kcal% protein and 34 kcal% lipids and comprises yogurt, cereals and almonds. Participants will be asked to consume the entire breakfast in less than 15 min and to complete a visual analog scale (VAS) questionnaire every 15 min. Blood sampling will be repeated at 60 min after starting breakfast (postprandial).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- food intake (breakfast) (Experimental): the breakfast composition is 56 kcal% carbohydrates, 12 kcal% protein and 34 kcal% lipids and comprises yogurt, cereals and almonds
  Interventions: Dietary Supplement: food (breakfast)

INTERVENTIONS:
Dietary Supplement: food (breakfast) — The breakfast composition is 56 kcal% carbohydrates, 12 kcal% protein and 34 kcal% lipids and comprises yogurt, cereals and almonds

SUMMARY:
The present study aims to evaluate in adults with normal weight and with overweight or obesity who live in the city of La Plata the circulating levels of various hormones that regulate appetite and the gene expression of their receptors in peripheral blood mononuclear cells before and after food intake.

DETAILED DESCRIPTION:
the investigators plan a single test meal study in males and females with normal weight (NW) or overweight/obesity (OW/OB) assessing whether plasma appetite regulatory hormones levels are associated with different metabolic and anthropometric variables as well as with appetite sensations.

ELIGIBILITY:
Inclusion Criteria:

* adult individuals body mass index> 18.5 kg∙m-2

Exclusion Criteria:

* chronic medical illness, personal history of diabetes, history of medical condition, or medication related to obesity or diabetes risk status.

Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
plasma ghrelin concentration | pre -prandial
  ghrelin concentration (fmol/ml)
plasma leptin concentration | pre -prandial
  leptin concentration (ug/ml)
plasma glucagon-like peptide 1 concentration | pre -prandial
  glucagon-like peptide 1 concentration (ug/ml)
plasma liver antimicrobial peptide 2 concentration | pre -prandial
  liver antimicrobial peptide 2 concentration (pmol/ml)
plasma des-acyl ghrelin concentration | pre -prandial
  des-acyl ghrelin concentration (fmol/ml)
plasma ghrelin concentration | 1 hour post -prandial
  ghrelin concentration (fmol/ml)
plasma leptin concentration | 1 hour post -prandial
  leptin concentration (ug/ml)
plasma glucagon-like peptide 1 concentration | 1 hour post -prandial
  glucagon-like peptide 1 concentration (ug/ml)
plasma liver antimicrobial peptide 2 concentration | 1 hour post -prandial
  liver antimicrobial peptide 2 concentration (pmol/ml)
plasma des-acyl ghrelin concentration | 1 hour post -prandial
  des-acyl ghrelin concentration (fmol/ml)
plasma glucose concentration | pre -prandial
  glucose concentration (mg%)
plasma glucose concentration | 1 hour post -prandial
  glucose concentration (mg%)
plasma triglycerides concentration | pre-prandial
  triglycerides concentration (mg%)
plasma triglycerides concentration | 1 hour post -prandial
  triglycerides concentration (mg%)
plasma total cholesterol concentration | pre -prandial
  total cholesterol concentration (mg%)
plasma total cholesterol concentration | 1 hour post -prandial
  total cholesterol concentration (mg%)
ghrelin proteolysis | pre -prandial
  plasma proteolytic activity of ghrelin (relative units)
ghrelin proteolysis | 1 hour post -prandial
  plasma proteolytic activity of ghrelin (relative units)
ghrelin deacylation | pre -prandial
  plasma desacylase actvitity of ghrelin (relative units)
ghrelin deacylation | 1 hour post -prandial
  plasma desacylase actvitity of ghrelin (relative units)
leptin receptor gene expression in peripheral blood mononuclear cells | pre-prandial
  leptin receptor gene expression in peripheral blood mononuclear cells (relative expression)
insulin receptor gene expression in peripheral blood mononuclear cells | pre-prandial
  insulin receptor gene expression in peripheral blood mononuclear cells (relative expression)
ghrelin receptor gene expression in peripheral blood mononuclear cells | pre-prandial
  ghrelin receptor gene expression in peripheral blood mononuclear cells (relative expression)
hunger sensation | pre-prandial and 15, 30, 45 and 60 min post-prandial
  visual analog scale (cm)
fullness sensation | pre-prandial and 15, 30, 45 and 60 min post-prandial
  visual analog scale (cm)
"desire to eat" sensation | pre-prandial and 15, 30, 45 and 60 min post-prandial
  visual analog scale (cm)
"prospective food consumption" sensation | pre-prandial and 15, 30, 45 and 60 min post-prandial
  visual analog scale (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Andreoli, Principal Investigator — Instituto de Desarrollo e Investigaciones Pediátricas (IDIP)
Locations (1):
- Instituto de Desarrollo e Investigaciones Pediátricas (IDIP), La Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andreoli MF, Fittipaldi AS, Castrogiovanni D, De Francesco PN, Valdivia S, Heredia F, Ribet-Travers C, Mendez I, Fasano MV, Schioth HB, Doi SA, Habib AM, Perello M. Pre-prandial plasma liver-expressed antimicrobial peptide 2 (LEAP2) concentration in humans is inversely associated with hunger sensation in a ghrelin independent manner. Eur J Nutr. 2024 Apr;63(3):751-762. doi: 10.1007/s00394-023-03304-8. Epub 2023 Dec 29. PMID 38157050